CLINICAL TRIAL: NCT05647278
Title: Tegoprazan-Amoxicillin Dual Therapy Versus Esomeprazole-Based Bismuth Quadruple Therapy for First-Line Helicobacter Pylori Eradication: A Prospective, Randomized, Multicenter, Superiority Study (TATH-1)
Brief Title: Tegoprazan-Amoxicillin Dual Therapy vs. Bismuth Quadruple Therapy for H. Pylori Infection (TATH-1)
Acronym: TATH-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhang Xiaofeng,MD (Other)
Responsible Party: Sponsor-Investigator, Zhang Xiaofeng,MD, chief physician, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-184
Record Dates: First submitted 2022-11-23; First posted 2022-12-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication
MeSH Terms: interventions — tegoprazan; Tablets; Esomeprazole; BID protein, human; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tegoprazan 50mg QD (Experimental): Tegoprazan 50 mg once daily plus Amoxicillin 1000mg TID for up to 2 weeks
  Interventions: Drug: Tegoprazan 50 mg, tablets, orally, qd; Drug: amoxicillin 1000mg tid
- Esomeprazole 20 mg BID (Active Comparator): esomeprazole 20 mg, tablets, orally, bid given in combination with amoxicillin 1000mg，clarithromycin 500mg bid，colloidal bismuth pectin 200mg bid for up to 2 weeks.
  OR esomeprazole 20 mg, tablets, orally, bis in die given in combination with amoxicillin 750mg capsules, orally, quarter die for up to 2 weeks.
  Interventions: Drug: Esomeprazole 20mg BID; Drug: amoxicillin +clarithromycin+colloidal bismuth pectin BID
- Tegoprazan 50 mg BID (Experimental): Tegoprazan 50 mg twice daily plus Amoxicillin plus Amoxicillin 1000mg TID for up to 2 weeks
  Interventions: Drug: Tegoprazan 50 mg, tablets, orally, bid; Drug: amoxicillin 1000mg tid

INTERVENTIONS:
Drug: Tegoprazan 50 mg, tablets, orally, qd — Tegoprazan 50 mg, tablets, orally, qd given in combination with amoxicillin 1000mg capsules, orally, tid for up to 2 weeks.
  Arms: Tegoprazan 50mg QD
Drug: Esomeprazole 20mg BID — esomeprazole 20 mg, tablets, orally, bid given in combination with amoxicillin 1000mg，clarithromycin 500mg bid，colloidal bismuth pectin 200mg bid for up to 2 weeks.
  OR esomeprazole 20 mg, tablets, orally, bis in die given in combination with amoxicillin 750mg capsules, orally, quarter die for up to 2 weeks.
  Arms: Esomeprazole 20 mg BID
Drug: Tegoprazan 50 mg, tablets, orally, bid — Tegoprazan 50 mg, tablets, orally, bid given in combination with amoxicillin 1000mg capsules, orally, tid for up to 2 weeks.
  Arms: Tegoprazan 50 mg BID
Drug: amoxicillin +clarithromycin+colloidal bismuth pectin BID — amoxicillin 1000mg，clarithromycin 500mg bid，colloidal bismuth pectin 200mg bid for up to 2 weeks
  Arms: Esomeprazole 20 mg BID
Drug: amoxicillin 1000mg tid — amoxicillin 1000mg tid
  Arms: Tegoprazan 50 mg BID; Tegoprazan 50mg QD

SUMMARY:
Standard eradication therapies using proton pump inhibitors (PPIs) require double doses to achieve sufficient acid suppression, yet failure rates remain high due to antibiotic resistance. Tegoprazan, a P-CAB agent, inhibits gastric acid more effectively than PPIs. This study hypothesizes that Tegoprazan-based dual therapy can achieve superior or non-inferior eradication rates compared to standard quadruple therapy. The study evaluates the antibacterial effect of Tegoprazan combined with high-dose Amoxicillin in H. pylori-infected patients.

DETAILED DESCRIPTION:
Note on Protocol Amendment and Registration Update: The study protocol was amended in November 2023 to include a randomized comparison of Tegoprazan 50 mg QD versus BID (within the TAT arm) and to adjust the Amoxicillin dosage to 1000 mg TID. Important Explanation: Although this amendment was approved by the Ethics Committee and implemented immediately, the update to the ClinicalTrials.gov registry was delayed due to an administrative oversight by the research team. The inclusion of the BID arm and the secondary randomization were pre-planned and executed strictly according to the protocol, not as a post-hoc analysis.

Study Description: Helicobacter pylori infection is a major cause of gastric diseases. Currently, Bismuth Quadruple Therapy (BQT) is the recommended first-line treatment in China. However, the efficacy of BQT is increasingly challenged by antibiotic resistance (especially to clarithromycin) and complex dosing regimens, which can reduce patient compliance.

Tegoprazan is a novel potassium-competitive acid blocker (P-CAB) that provides rapid, potent, and durable acid suppression, theoretically creating an ideal environment for amoxicillin to eradicate H. pylori. Unlike proton pump inhibitors (PPIs), Tegoprazan does not require activation by acid and is less influenced by CYP2C19 genetic polymorphisms.

This prospective, randomized, multicenter study aims to compare the efficacy, safety, and compliance of 14-day Tegoprazan-Amoxicillin Dual Therapy (TAT) versus Esomeprazole-based Bismuth Quadruple Therapy (BQT) in treatment-naïve patients. The study hypothesizes that the TAT regimen is superior or non-inferior to the standard BQT regimen in eradicating H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years with Hp-positive first sterilization were included in this study.
2. Before treatment, the existence of Helicobacter pylori can be confirmed by one or more of the following methods: rapid urease test, Hp culture, 13C urea breath test, 14C urea breath test and stool Hp antigen test.

Exclusion Criteria:

1. acute upper gastrointestinal bleeding.
2. active gastric or duodenal ulcer.
3. acute gastric or duodenal mucosal lesions.
4. previous eradication treatment of Helicobacter pylori.
5. penicillin/furazolidone allergy.
6. surgery that may affect gastric acid secretion (upper gastrointestinal resection or vagotomy).
7. Zollinger-Ellison syndrome or other hypergastric acid secretion diseases.
8. severe neurological, cardiovascular, pulmonary, liver,renal, metabolic,gastrointestinal, urological, etc.
9. Any fertile woman must use proper contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Helicobacter Pylori Positive (HP+) Participants With Successful HP Eradication at Week 4 Post- Treatment | Week 4-8 post-treatment
  HP infection status will be determined by ^13C Urea Breath Test (^13C-UBT). The urea breath test is used to detect infection with HP, a bacteria associated with stomach ulcers, by testing individual breath samples in a central laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou first people's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No